CLINICAL TRIAL: NCT04763512
Title: Clinical Study of Partially Hydrolysed Protein Infant Formula on Trans-epidermal Water Loss (TEWL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Medidata Solutions (Industry); SAS Institute (Industry); Veeva Systems (Industry); Cognizant Technology Solutions AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20.16.INF
Record Dates: First submitted 2020-11-19; First posted 2021-02-21 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis; Skin Condition
Keywords: atopic dermatitis development; trans-epidermal water loss; allergy; growth patterns; quality of life; gut comfort; partially hydrolysed whey
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intact Cow's Milk Protein Formula Group (CMFG) (Experimental): All enrolled subjects will be fed Stage 1 CMF libitum for 4 months. Thereafter, they will discontinue study formula and complete the study.
  Interventions: Dietary Supplement: Intact Cow's Milk Protein Formula
- Partially Hydrolysed Whey Formula Group (pHFG) (Experimental): All enrolled subjects will be fed Stage 1 pHF libitum for 4 months. Thereafter, they will switch to Stage 2 pHF at age 6 months (Study Month 4) and to Stage 3 pHF at age 12 months (Study Month 9) and continue until age 18 months (Study Month 15). Thereafter, they will discontinue study formula and complete the study.
  Interventions: Dietary Supplement: Partially Hydrolysed Whey Formula

INTERVENTIONS:
Dietary Supplement: Intact Cow's Milk Protein Formula — Study product will be provided as powder, reconstituted with water by parents/caregivers according to label instructions, and consumed orally. Study participants will continue this feeding regimen for 4 months.
  Arms: Intact Cow's Milk Protein Formula Group (CMFG)
Dietary Supplement: Partially Hydrolysed Whey Formula — Study product will be provided as powder, reconstituted with water by parents/caregivers according to label instructions, and consumed orally. Study participants will continue this feeding regimen for 16 months.
  Arms: Partially Hydrolysed Whey Formula Group (pHFG)

SUMMARY:
This is a single-centre, prospective, randomized, open-label, controlled trial of 200 infants 42±7 days of age. Subjects will be randomized to one of two open label feeding intervention group:

* Intact Cow's Milk Protein Formula Group (CMFG) (n = 100) or
* Partially Hydrolysed Whey Formula Group (pHFG) (n = 100).

DETAILED DESCRIPTION:
Atopic dermatitis (AD) affects 15 - 30% of children. Approximately 45% of these cases have an onset within the first 6 months of life and 60% develop within the first year (Bieber 2010). Besides environmental factors, the aetiology of AD has been found to be associated with genetic variants involved in skin barrier function defect and inflammation, leading to dry skin with increases in susceptibility to environmental exposures (Bieber 2008).

Partially hydrolysed cow's milk (whey) protein infant formula (pHF) has been shown to be effective in prevention of AD, both among at-risk and healthy infants (Exl, Deland et al. 2000, von Berg, Koletzko et al. 2003, Jingrana and Dunjina 2015). However, to date there are no published pediatric data to document the relationship between partially hydrolysed protein formulas and skin barrier function, specifically evaluating the effect of pHF on Trans-epidermal Water Loss (TEWL) among infants. Therefore, this study aims to evaluate the effect on skin barrier function as measured by TEWL and we hypothesize that infants consuming partially hydrolysed starter formula will have lower TEWL when compared infants consuming intact cow's milk protein starter formula.

ELIGIBILITY:
Inclusion Criteria:

* Infants 42± 7 days of age at enrolment (date of birth = age 0).
* Infants who have been born full-term gestational birth (≥ 37 completed weeks of gestation) and having a birth weight ≥ 2.5 kg and ≤ 4.5 kg.
* Parents /caregivers must agree to follow study procedures and recommended skincare routines, such as avoidance of moisturizers or other skincare products on the primary sites of interest.
* Parent(s) must have already independently elected before enrolment to formula feed and less than 30% of intake will be from breastmilk.

Exclusion Criteria:

* Known and diagnosed cow's milk protein allergy/intolerance.
* Infants currently using or have ever used partially hydrolysed protein formulas.
* Infants who have ever used topical corticosteroids, calcineurin inhibitors and/or any other physician-recommended treatments for skin conditions after birth.
* Infants who have been introduced to complementary foods.

Ages: 35 Days to 49 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Skin barrier function | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months)
  Change in Trans-epidermal water loss (TEWL)

SECONDARY OUTCOMES:
Weight | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Weight in grams and corresponding Z-score according to WHO reference standards and/or local standardized growth charts will be calculated.
Length | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Length in centimeters and corresponding Z-score according to WHO reference standards and/or local standardized growth charts will be calculated.
Head Circumference | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Head circumference in centimeters and corresponding Z-score according to WHO reference standards and/or local standardized growth charts will be calculated.
Infant health-related quality of life | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Assessed through a parent-reported, validated questionnaire called Infant Toddler Quality of Life questionnaire 47-item short-form (ITQOL-SF47). For each concept, item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health).
Infant health-related quality of life | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Assessed through the Happy Growth Index Questionnaire with each question rated on a Likert scale from strongly disagree to strongly agree.
Incidence and severity of Atopic Dermatitis (AD) and other allergic manifestations (CMF group) | aseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Incidence will be gathered from standard Adverse Event (AE) reporting. Atopic Dermatitis (AD) will be diagnose based on the Williams diagnostic criteria of International Study of Asthma and Allergies in Childhood (ISAAC). Severity of AD will be assessed using the SCORing Atopic Dermatitis (SCORAD) index, which consists of the extent and intensity of the disorder and subjective symptoms.
Infant gut comfort | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months)
  Using the Infant Gastrointestinal Symptom Questionnaire (IGSQ)-13.
Toddler gut comfort | Study Month 9 (age 12 months) and Study Month 15 (age 18 months)
  Using the Toddler Gut Comfort Questionnaire.
Stool consistency | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months)
  Parents will record for 3 consecutive days after each bowel movement in a 3-Day Stool Diary the stool consistency on a validated 5-point scale from 1-watery to 5-hard.
Formula acceptance and satisfaction | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Formula intake, acceptability and satisfaction recorded using the Milk Intake and Satisfaction Questionnaire.
Safety assessment: Adverse events (AEs) | Baseline (age 42 ± 7 days) to Study Month 4 (age 6 months) - in both randomized groups and until Study Month 15 (age 18 months) in pHF group only
  Using standard adverse events (AEs) reporting for safety assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Shao, Dr., Principal Investigator — Shanghai Tonxin Pediatric Clinic Co. Ltd
Locations (1):
- Shanghai Tonxin Pediatric Clinic Co. Ltd, Shanghai, Shanghai Municipality, China